CLINICAL TRIAL: NCT02229006
Title: SoFIA3: Sodium Fluoride Imaging (18F-NaF PET-CT) in Abdominal Aortic Aneurysms
Brief Title: Sodium Fluoride Imaging of Abdominal Aortic Aneurysms
Acronym: SoFIA3
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Other Study IDs: ETM/365
Record Dates: First submitted 2014-08-25; First posted 2014-08-29 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2016-10

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Aortic aneurysm, abdominal; Sodium Fluoride; Positron Emission Tomography
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aneurysm surveillance: Radiation: 18F-NaF PET-CT
  Interventions: Radiation: 18F-NaF PET-CT
- Control patients: Radiation: 18F-NaF PET-CT
  Interventions: Radiation: 18F-NaF PET-CT

INTERVENTIONS:
Radiation: 18F-NaF PET-CT

SUMMARY:
The purpose of this study is to determine whether Sodium Fluoride imaging (using Positron Emission Tomography-Computed Tomography - PET-CT) is able to help predict the rate of abdominal aortic aneurysm expansion.

DETAILED DESCRIPTION:
Ruptured abdominal aortic aneurysms (AAAs) have a 90% mortality rate but there are currently no accurate methods of establishing the risk of rupture for an individual patient with an asymptomatic AAA. In vascular disease, microcalcification occurs in response to necrotic inflammation. Using computed tomography and positron emission tomography (PET-CT), early micro calcification can be identified using uptake of the radiotracer 18F-sodium fluoride. This can identify high risk-lesions in the aorta, coronary and carotid arteries, and appears to be indicative of necrotic and heavily inflamed tissue. The study investigators therefore propose to evaluate the ability of 18F-sodium fluoride to identify regions of necrotic inflammation in AAA and predict AAA expansion. The study investigators will explore its value as part of an ongoing clinical trial assessing the identification of macrophage activity using magnetic resonance imaging - the MA3RS Study (ISRCTN76413758). Patients already enrolled in the MA3RS Study will be recruited for the SoFIA3 study. Control patients with a normal calibre aorta will be recruited from the National AAA Screening Programme.

ELIGIBILITY:
Inclusion Criteria (AAA patients):

* Patients already enrolled in the MA3RS study (ISRCTN76413758)
* Patients with abdominal aortic aneurysm with AP diameter >40 mm on ultrasound
* >50 years of age

Inclusion Criteria (control patients):

* Patients with abdominal aorta with AP diameter <30 mm on ultrasound
* >50 years of age

Exclusion Criteria:

* Patients expected to undergo imminent AAA repair
* Patients who refuse or are unable to give informed consent
* Women of child-bearing potential without contraception
* Patients who are unable to undergo PET-CT scan
* Patients with collagen vascular disease
* Intercurrent illness, malignancy or comorbidity with life expectancy <1 year
* Renal dysfunction (eGFR <30ml/min/1.73m2)
* Contraindication to PET-CT or CTA
* Iodine allergy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case: patients with abdominal aortic aneurysm enrolled in the hospital ultrasound surveillance programme Control: patients with normal calibre aorta as demonstrated from an ultrasound performed as part of the National AAA Screening Programme
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2014-09; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in abdominal aortic aneurysm anteroposterior diameter over time at 6 and 12 months (mm) | 0, 6, 12 months
  The maximum AAA AP diameter on ultrasound will be obtained from time points below:
  1. At (or close to) the time of the study visit
  2. 6 months following the study visit
  3. 12 months following the study visit
  The maximum AP diameter will also be recorded on CTA performed at the time of study visit.

SECONDARY OUTCOMES:
Co-localisation of 18F-NaF with USPIO uptake on MRI scanning | At baseline
  The data on USPIO uptake on MRI scanning will be derived from a separate study (MA3RS - MRI in AAA to predict Rupture or Survival, ISRCTN76413758). The proposed study described here (SoFIA3) will not involve any administration of USPIO.
  Regions of interest and uptake of 18F-NaF will be identified on PET-CT images acquired at baseline as part of this study (SoFIA3). These images will be co-registered to MRI data (uptake pre- and post-USPIO) which has already been obtained during the MA3RS Study. We will correlate the agreement between areas of significant 18F-NaF uptake on PET-CT (representing areas of active calcification) and areas of significant USPIO uptake on MRI (representing areas of active macrophage activity).
  This is an exploratory analysis which will take advantage of data already obtained through the MA3RS Study, which is a separate study.

OTHER OUTCOMES:
Co-localisation of 18F-NaF with histological evidence of active calcification, necrotic inflammation and proteolytic degradation of the aneurysm wall | At baseline
  Uptake of 18F-NaF will be identified on PET-CT scans that are acquired as part of the study visit. We will take advantage of histological tissue specimens that will be collected as part of the separate MA3RS Study (patients enrolled in the MA3RS Study who undergo AAA repair give consent to tissue samples being take and analysed).
  We will take advantage of histological data that is already obtained from the MA3RS study and use this to correlate histological areas of inflammation with areas of active calcification on PET-CT.
Relationship with areas of high wall stress (finite element analysis) | At baseline
  As part of the MA3RS Study, patients will undergo CTA scans at baseline and 24 months. These are being used by other members of the team in the development of novel imaging techniques to quantify areas of high wall stress, through finite element analysis.
  The extra CTA and calcium scoring scans acquired as part of SoFIA3 (which could be at any time following the first MA3RS CTA) may contribute to this image analysis technique.
Comparison of 18F-NaF uptake in patients with AAA versus control patients | At baseline
  We will compare objective measures of tracer uptake in AAA vs control aorta

CONTACTS AND LOCATIONS:
Overall Officials: Rachael O Forsythe, MD, Principal Investigator — University of Edinburgh; David E Newby, MD PhD, Study Director — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Debono S, Tzolos E, Syed MBJ, Nash J, Fletcher AJ, Dweck MR, Newby DE, Dey D, Forsythe RO, Williams MC. CT Attenuation of Periaortic Adipose Tissue in Abdominal Aortic Aneurysms. Radiol Cardiothorac Imaging. 2024 Feb;6(1):e230250. doi: 10.1148/ryct.230250. PMID 38329405
- [Derived] Forsythe RO, Dweck MR, McBride OMB, Vesey AT, Semple SI, Shah ASV, Adamson PD, Wallace WA, Kaczynski J, Ho W, van Beek EJR, Gray CD, Fletcher A, Lucatelli C, Marin A, Burns P, Tambyraja A, Chalmers RTA, Weir G, Mitchard N, Tavares A, Robson JMJ, Newby DE. 18F-Sodium Fluoride Uptake in Abdominal Aortic Aneurysms: The SoFIA3 Study. J Am Coll Cardiol. 2018 Feb 6;71(5):513-523. doi: 10.1016/j.jacc.2017.11.053. PMID 29406857